CLINICAL TRIAL: NCT01114776
Title: Pilot Study Examining Mechanisms of Iron Trafficking and Extra-hepatic Iron Distribution in Sickle Cell Disease, Thalassemia, and Other Iron Loading Anemias
Brief Title: Multi-Center Study of Iron Overload: Pilot Study
Acronym: MCSIO
Status: Completed | Type: Observational
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University College London (UCL) Cancer Institute (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Medical University Innsbruck (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-068; R01DK057778-06A1 (NIH)
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Sickle Cell Disease; Thalassemia; Diamond-Blackfan Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia, Diamond-Blackfan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Sickle Cell Disease (SCD): Patients with sickle cell diseases, 16 years or older with 10-20 years of transfusion (defined as 0.2-0.6mg Fe/kg/day exposure with annual ferritin levels greater than 2500 in at least 60% of years of chronic transfusion); 0 to 9 years old at the initiation of chronic transfusions; no exchange transfusions in the previous 6 months; and iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months or ferritin level greater than 1500mg/dl.
- Thalassemia Major (TM): Patients with β-thalassemia major and transfusion-dependent E-beta THAL. 16 years or older with 10-20 years of chronic transfusion (defined above), 0 to 9 years old at the initiation of chronic transfusions, iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months.
- Diamond Blackfan Anemia (DBA): Patients with DBA, 16 years or older with 10-20 years of transfusion, 0 to 9 years old at the initiation of chronic transfusions, iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months.
- Controls

SUMMARY:
The purpose of this study is to initiate pilot studies to demonstrate that a sufficient number of iron-overloaded thalassemia, SCD and DBA populations with similar duration of chronic transfusion, and age at start of transfusions would be available for a confirmatory study and to validate that proposed multicenter MRI and biochemical studies can be completed. The study will examine the hypothesis that a chronic inflammatory state in Sickle Cell Disease (SCD) leads to hepcidin- and cytokine-mediated iron withholding within the RES (reticuloendothelial system), lower plasma NTBI (non transferrin bound iron) levels, less distribution of iron to the heart in SCD.

DETAILED DESCRIPTION:
A detailed iron burden, transfusion and chelation history will be obtained from chart review or from participant recall.

Iron burden data will include: 1) documentation of liver iron, and 2) average annual ferritin values.

Transfusion data will include: (1) age at onset of regular transfusions, (2) years of chronic transfusion therapy, and (3) pre-transfusion Hb calculated as average of all assessments for each year.

MRI will be performed measuring pituitary, cardiac, and liver iron.

Laboratory samples should be obtained pre-transfusion and mid-cycle.

All interviews, exams, laboratory tests, study procedures and MRI assessments should be completed within a 0 to 12 weeks time span.

In addition, a healthy control group will also be recruited with similar age, gender, and ethnicity as the disease groups.

ELIGIBILITY:
Inclusion Criteria:

* 10-20 years of transfusion (defined as 0.2-0.6mg Fe/kg/day exposure with annual ferritin levels greater than 2500 in at least 60% of years of chronic transfusion);
* 0 to 9 years old at the initiation of chronic transfusions; no exchange transfusions in the previous 6 months
* iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months or ferritin level greater than 1500mg/dl.

Exclusion Criteria:

* Patients with HbSC, HbS/β thalassemia
* Pacemaker (active or inactive) or other implanted magnetic devices, severe claustrophobia, or other contraindications to MRI; Unable to remove ferro-magnetic objects from the body in regions to be imaged (e.g., jewelry or piercing)
* Presence of any other condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment;
* Any chronic inflammatory illness other than the SCD, TM or DBA;
* Any acute illness within a 14 day period prior to blood sampling;
* Patients receiving intensive chelation in the 6 months prior to enrollment including deferoxamine 24 hours per day, 7 days per week or combination treatment with 2 chelators
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There is no gender predisposition for sickle cell disease, thalassemia major, or Diamond-Blackfan anemia. Sickle cell anemia most frequently affects people of African descent, thalassemia affects people of Mediterranian, northern African, Southeast Asia and Indian descent. Diamond-Blackfan anemia occurs across all racial and ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11-01; Primary Completion 2013-07-31 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Pilot study of biochemical mechanisms of iron deposition in patients with Sickle Cell Disease, Thalassemia and Diamond-Blackfan Anemia. | March 2010 - August 2012
  To examine the hypothesis that a chronic inflammatory state in Sickle Cell Disease (SCD) leads to hepcidin- and cytokine-mediated iron withholding within the RES (reticuloendothelial system), lower plasma NTBI (non transferrin bound iron) levels, less distribution of iron to the heart in SCD, and finally lower uptake and enhanced export of NTBI by cardiomyocytes conditioned by SCD serum, when compared with similarly iron overloaded patients with beta thalassemia and diamond blackfan anemia.

SECONDARY OUTCOMES:
Comparison of cardiac and pituitary iron content by MRI | March 2010 - August 2012
  We will measure cardiac and pituitary iron deposition by MRI in SCD with 10-20 years of transfusion exposure (0.2-0.6 mg Fe/kg/day) and compare this to measurements in a similarly transfused group of TM (or DBA). Patients with similar duration of chronic transfusion and age at onset of chronic transfusion therapy will be compared.
Characterization of levels and speciation of NTBI in heavily transfused SCD vs. TM (or DBA) | March 2010 - August 2012
  Levels of total and speciated NTBI (directly chelatable, labile plasma (LPI) and bleomycin-reactive) will be correlated with inflammatory biomarkers, hepcidin levels and organ iron deposition in patients with SCD, TM (or DBA). Results from the 3 patient populations will be compared to determine the possible effect of ineffective erythropoiesis in TM on the amount or species of NTBI present in the circulation.
To examine mediators of iron trafficking including inflammatory and regulatory cytokines (TNF-α, IL-1, IL-6, IL-10, TGF β), hepcidin, and nutritional factors (Vitamin C and D) in heavily transfused patients with SCD and TM (or DBA) | March 2010 - August 2012
  To examine the hypothesis that disease-related differences in inflammatory markers, hepcidin, and nutritional factors affect NTBI deposition, we will define the relationships between plasma and monocyte cytokines known to have cellular effects on iron cell trafficking (IL-1, IL-6, IL-10, TNFalpha, and TGFbeta), hepcidin concentration, and nutrient factors on NTBI levels and characteristics.
To examine the cellular mechanisms of iron sequestration in the RES and uptake of iron into other iron storage sites in SCD relative to TM (or DBA) | March 2010 - August 2012
  We will examine iron homeostasis in primary monocytes obtained from the 4 study groups to ascertain whether there is increased iron accumulation in monocytes in SCD patients. We will determine total cellular iron and ferritin-bound iron in monocytes isolated from the blood of SCD, TM and DBA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; John B Porter, MD, Principal Investigator — University College London (UCL) Cancer Institute
Locations (3):
- Children's Hospital & Research Center Oakland, Oakland, California, United States
- Universitätsklinikum Hamburg-Eppendorf, Hamburg-Eppendorf, Germany
- UCL Cancer Institute, London, United Kingdom